CLINICAL TRIAL: NCT06823739
Title: Personalized Diet with or Without Physical Exercise Improves Nutritional Status, Muscle Strength, Physical Performance and Quality of Life in Malnourished Older Adult Patients: a Prospec-tive Randomized Controlled Study
Brief Title: Personalized Diet and Physical Exercise in Malnourished Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Mustafa Altınkaynak, associate professor, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 228630-2021
Record Dates: First submitted 2025-02-05; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Malnourished Elderly; Quality of Life (QOL); BMI; Hand Grip Strength; Timed Up and Go
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- personalized diet (No Intervention): Participants in this group received an individualized nutritional intervention tailored to their energy and protein needs (25-30 kcal/kg/day and 1.0-1.2 g/kg/day, respectively). The diet plan included a balance of macronutrients (45-55% carbohydrates, 20-35% fats, and 20-30 g fiber daily) and emphasized protein diversity, whole grains, healthy fats, and adequate hydration. Weekly phone calls monitored adherence to the diet.
- Personalized Diet with Physical Exercise (Active Comparator): Participants in this group received the same personalized diet intervention as the PD group, but with the addition of a structured home-based physical exercise program. The program included:
  Warm-up (10 min): Stretching, posture exercises, and stationary marching Strength and balance training (20 min): Bodyweight exercises, balance drills, and brisk walking (10-30 min per session) Cool-down (10 min): Gentle stretching and relaxation
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — This exercise program in PDE group was designed to be performed at home without re-quiring any specialized equipment. It aims to improve physical health, balance, and coor-dination while maintaining muscle strength and flexibility. Patients performed brist walking at least three times a week for a duration of 10 to 30 minutes per session. It also included balance practice and coordination exercises for 10 minutes. These include: Standing on tiptoes, balancing on one foot while holding onto a chair for support, walking in a straight line as if on a narrow beam. Finally, the exercise session ended with a 10-minute cool-down, focusing on relaxing muscles and performing gentle stretches to improve flexibility and reduce tension. All of the exercises were both explained and given in a figured chart, to the patients or the relatives
  Arms: Personalized Diet with Physical Exercise

SUMMARY:
In this study, personalized diet therapy will be planned by expert dietitians for the volunteers, and they will be instructed on simple stretching and strengthening exercises they can perform independently at home. This instruction will also be supported visually.

During the study, the body composition of the volunteers (muscle mass and percentage, fat mass and percentage) will be measured using a BIA device, and their height and weight will also be recorded. Hand grip strength will be measured using a device called a dynamometer.

These measurements will be repeated monthly for a total of 3 months.

To assess the quality of life of the volunteers, a questionnaire-based test will be conducted, and these measurements will also be repeated monthly for 3 months.

Furthermore, the physical performance of the volunteers will be evaluated by having them stand up from a chair, walk 3 meters, return, and sit back down. This duration will be measured in seconds and recorded. These measurements will also be repeated monthly for 3 months.

Volunteers have no obligations in this research.

Since no invasive procedures (e.g., incisions, tissue or blood sampling, or use of medical devices to examine internal parts of the body) or medical drug therapies will be applied, the risks to the volunteers are minimal.

By implementing personalized diets and standard physical exercise programs, it is anticipated that volunteers will receive medical benefits.

Participation in the study is voluntary, and volunteers can refuse to participate or withdraw from the study at any time without facing any penalties or sanctions and without losing any rights.

Observers, auditors, the ethics committee, institutions, and other relevant health authorities may have direct access to the medical records of the volunteers. However, this information will be kept confidential. By signing this informed consent form, the volunteer and their legal representative grant permission for such access.

Records that reveal the identity of the volunteer will be kept confidential in accordance with relevant regulations, will not be disclosed to the public, and the identity of the volunteer will remain confidential even if the research results are published.

If new information is obtained during the research that could affect the willingness of the volunteer to continue participating, the volunteer and their legal representative will be informed promptly.

For information about the research, the volunteer's rights, or any adverse events related to the research, the volunteer can contact the individuals listed below 24/7 using the provided contact details.

The anticipated duration for a volunteer to participate in this research is 3 months.

No biological material will be obtained from volunteers in this research.

ELIGIBILITY:
Inclusion Criteria:

* Malnourished old aged patients (≥65 years old) who were oriented, cooperated, and inde-pendent in daily living activities were included in the study

Exclusion Criteria:

* Exclusion criteria were; <65 years of age, cognitive impairment, immobilization, eat-ing/swallowing disorders, receiving enteral or parenteral nutritional support, and having acute medical problems.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes — over aged 65
Enrollment: 20 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Improvement in Nutritional Status, Muscle Strength, Quality of Life and Physical Performance in Malnourished Older Adults | Baseline, 4th week, 8th week, and 12th week
  The Mini Nutritional Assessment--Short Form (MNA-SF) test was performed . Body mass index (BMI) was calculated by body weight (kg) by square of the body height (m), and is expressed in kg/m2. The appendicular skeletal muscle mass (ASM) was measured through BIA using a Tanita MC 780 MA (Japan). The ASM index (ASMI) was calculated with by dividing the ASM by the square of the body height (kg/m2).
  Muscle strength was measured using a standardized handheld dynamometer (Jamar, USA), the best of 3 measurements made the dominant hand.
  A TUG test was performed to evaluate physical performance. The patients sat on a standard chair and were then told to get up from the chair, walk to a line 3 meters away, come back, and sit on the chair again.
  The EuroQoL-5 Dimensions (EQ-5D) quality-of-life score and visual analog scale (EQ-5D VAS) were used to assess quality of life. The index score ranged from -0.59 to 1. -0.59 indicates a quality of life worse than death and 1 is a perfect life quality

SECONDARY OUTCOMES:
Correlation between the QoL score and Body Mass Index, Mını Nutritional Assessment Short Form, Hand Grip Strength, Appendiculer Muscle Mass Index, Timed up and Go | 0th and 12th weeks
  Correlation between the QoL score and other variables' changes are calculated after 12 weeks of intervention in the whole study group with Spearman correlations

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Faculty of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Background] Lu X, Chu H, Wang L, Yang R, Li Y, Sun W, Yan C, Liu Y, Guo Z, Cheng X. Age- and sex-related differences in muscle strength and physical performance in older Chinese. Aging Clin Exp Res. 2020 May;32(5):877-883. doi: 10.1007/s40520-019-01263-x. Epub 2019 Jul 2. PMID 31267378
- [Background] Groessl EJ, Kaplan RM, Barrett-Connor E, Ganiats TG. Body mass index and quality of well-being in a community of older adults. Am J Prev Med. 2004 Feb;26(2):126-9. doi: 10.1016/j.amepre.2003.10.007. PMID 14751323
- [Background] Nascimento MM, Gouveia ER, Gouveia BR, Marques A, Campos P, Garcia-Mayor J, Przednowek K, Ihle A. The Mediating Role of Physical Activity and Physical Function in the Association between Body Mass Index and Health-Related Quality of Life: A Population-Based Study with Older Adults. Int J Environ Res Public Health. 2022 Oct 22;19(21):13718. doi: 10.3390/ijerph192113718. PMID 36360598
- [Background] Ramsey KA, Meskers CGM, Trappenburg MC, Verlaan S, Reijnierse EM, Whittaker AC, Maier AB. Malnutrition is associated with dynamic physical performance. Aging Clin Exp Res. 2020 Jun;32(6):1085-1092. doi: 10.1007/s40520-019-01295-3. Epub 2019 Aug 19. PMID 31429000
- [Background] Steffen TM, Hacker TA, Mollinger L. Age- and gender-related test performance in community-dwelling elderly people: Six-Minute Walk Test, Berg Balance Scale, Timed Up & Go Test, and gait speeds. Phys Ther. 2002 Feb;82(2):128-37. doi: 10.1093/ptj/82.2.128. PMID 11856064
- [Background] Strasser B, Grote V, Bily W, Nics H, Riedl P, Jira I, Fischer MJ. Short-Term Effects of Dietary Protein Supplementation on Physical Recovery in Older Patients at Risk of Malnutrition during Inpatient Rehabilitation: A Pilot, Randomized, Controlled Trial. Healthcare (Basel). 2023 Aug 17;11(16):2317. doi: 10.3390/healthcare11162317. PMID 37628515
- [Background] Chew STH, Tan NC, Cheong M, Oliver J, Baggs G, Choe Y, How CH, Chow WL, Tan CYL, Kwan SC, Husain FS, Low YL, Huynh DTT, Tey SL. Impact of specialized oral nutritional supplement on clinical, nutritional, and functional outcomes: A randomized, placebo-controlled trial in community-dwelling older adults at risk of malnutrition. Clin Nutr. 2021 Apr;40(4):1879-1892. doi: 10.1016/j.clnu.2020.10.015. Epub 2020 Oct 15. PMID 33268143
- [Background] Labott BK, Bucht H, Morat M, Morat T, Donath L. Effects of Exercise Training on Handgrip Strength in Older Adults: A Meta-Analytical Review. Gerontology. 2019;65(6):686-698. doi: 10.1159/000501203. Epub 2019 Sep 9. PMID 31499496
- [Background] Abizanda P, Lopez MD, Garcia VP, Estrella Jde D, da Silva Gonzalez A, Vilardell NB, Torres KA. Effects of an Oral Nutritional Supplementation Plus Physical Exercise Intervention on the Physical Function, Nutritional Status, and Quality of Life in Frail Institutionalized Older Adults: The ACTIVNES Study. J Am Med Dir Assoc. 2015 May 1;16(5):439.e9-439.e16. doi: 10.1016/j.jamda.2015.02.005. Epub 2015 Apr 2. PMID 25841327
- [Background] Kramer CS, Groenendijk I, Beers S, Wijnen HH, van de Rest O, de Groot LCPGM. The Association between Malnutrition and Physical Performance in Older Adults: A Systematic Review and Meta-Analysis of Observational Studies. Curr Dev Nutr. 2022 Jan 29;6(4):nzac007. doi: 10.1093/cdn/nzac007. eCollection 2022 Apr. PMID 35415390
- [Background] Jiang M, Zou Y, Xin Q, Cai Y, Wang Y, Qin X, Ma D. Dose-response relationship between body mass index and risks of all-cause mortality and disability among the elderly: A systematic review and meta-analysis. Clin Nutr. 2019 Aug;38(4):1511-1523. doi: 10.1016/j.clnu.2018.07.021. Epub 2018 Jul 26. PMID 30082166
- [Background] Magzal F, Turroni S, Fabbrini M, Barone M, Vitman Schorr A, Ofran A, Tamir S. A personalized diet intervention improves depression symptoms and changes microbiota and metabolite profiles among community-dwelling older adults. Front Nutr. 2023 Sep 14;10:1234549. doi: 10.3389/fnut.2023.1234549. eCollection 2023. PMID 37794974
- [Background] Ordovas JM, Berciano S. Personalized nutrition and healthy aging. Nutr Rev. 2020 Dec 1;78(12 Suppl 2):58-65. doi: 10.1093/nutrit/nuaa102. PMID 33259626
- [Background] Cederholm T, Barazzoni R, Austin P, Ballmer P, Biolo G, Bischoff SC, Compher C, Correia I, Higashiguchi T, Holst M, Jensen GL, Malone A, Muscaritoli M, Nyulasi I, Pirlich M, Rothenberg E, Schindler K, Schneider SM, de van der Schueren MA, Sieber C, Valentini L, Yu JC, Van Gossum A, Singer P. ESPEN guidelines on definitions and terminology of clinical nutrition. Clin Nutr. 2017 Feb;36(1):49-64. doi: 10.1016/j.clnu.2016.09.004. Epub 2016 Sep 14. PMID 27642056
- [Background] Seid AM, Fentahun N. Prevalence of malnutrition among old people in Africa: systematic review and meta-analysis. BMJ Open. 2022 Nov 30;12(11):e065197. doi: 10.1136/bmjopen-2022-065197. PMID 36450428
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] Borg GA. Psychophysical bases of perceived exertion. Med Sci Sports Exerc. 1982;14(5):377-81. PMID 7154893
- [Background] Dorrington N, Fallaize R, Hobbs DA, Weech M, Lovegrove JA. A Review of Nutritional Requirements of Adults Aged >/=65 Years in the UK. J Nutr. 2020 Sep 1;150(9):2245-2256. doi: 10.1093/jn/nxaa153. PMID 32510125
- [Background] Volkert D, Beck AM, Cederholm T, Cruz-Jentoft A, Hooper L, Kiesswetter E, Maggio M, Raynaud-Simon A, Sieber C, Sobotka L, van Asselt D, Wirth R, Bischoff SC. ESPEN practical guideline: Clinical nutrition and hydration in geriatrics. Clin Nutr. 2022 Apr;41(4):958-989. doi: 10.1016/j.clnu.2022.01.024. Epub 2022 Mar 5. PMID 35306388
- [Background] Bischoff HA, Stahelin HB, Monsch AU, Iversen MD, Weyh A, von Dechend M, Akos R, Conzelmann M, Dick W, Theiler R. Identifying a cut-off point for normal mobility: a comparison of the timed 'up and go' test in community-dwelling and institutionalised elderly women. Age Ageing. 2003 May;32(3):315-20. doi: 10.1093/ageing/32.3.315. PMID 12720619
- [Background] Bahat G, Aydin CO, Tufan A, Karan MA, Cruz-Jentoft AJ. Muscle strength cutoff values calculated from the young reference population to evaluate sarcopenia in Turkish population. Aging Clin Exp Res. 2021 Oct;33(10):2879-2882. doi: 10.1007/s40520-021-01785-3. Epub 2021 Jan 27. PMID 33501623
- [Background] Lafzi N, Altinkaynak M, Goksoy Y, Tor YB, Akpinar TS, Erten SN, Saka B. Estimation of the appendicular skeletal muscle mass and phase angle cut-off values from a young Turkish reference population using multifrequency bioelectrical impedance analysis. Eur Rev Med Pharmacol Sci. 2024 Feb;28(4):1282-1288. doi: 10.26355/eurrev_202402_35449. PMID 38436161
- [Background] Tucker E, Luscombe-Marsh N, Ambrosi C, Lushington K. Nutritional status and quality-of-life of older adults in aged care: A systematic review and meta-analysis. Exp Gerontol. 2022 Jun 1;162:111764. doi: 10.1016/j.exger.2022.111764. Epub 2022 Mar 7. PMID 35271944
- [Background] Huynh NTH, Nguyen TTT, Pham HKT, Huynh NTH, Nguyen NT, Cao NT, Dung DV. Malnutrition, Frailty, and Health-Related Quality of Life Among Rural Older Adults in Vietnam: A Cross-Sectional Study. Clin Interv Aging. 2023 Apr 26;18:677-688. doi: 10.2147/CIA.S405847. eCollection 2023. PMID 37138949
- [Background] Tanski W, Wojciga J, Jankowska-Polanska B. Association between Malnutrition and Quality of Life in Elderly Patients with Rheumatoid Arthritis. Nutrients. 2021 Apr 12;13(4):1259. doi: 10.3390/nu13041259. PMID 33921207
- [Background] Rasheed S, Woods RT. Malnutrition and quality of life in older people: a systematic review and meta-analysis. Ageing Res Rev. 2013 Mar;12(2):561-6. doi: 10.1016/j.arr.2012.11.003. Epub 2012 Dec 8. PMID 23228882
- [Background] Katsas K, Mamalaki E, Kontogianni MD, Anastasiou CA, Kosmidis MH, Varlamis I, Hadjigeorgiou GM, Dardiotis E, Sakka P, Scarmeas N, Yannakoulia M. Malnutrition in older adults: Correlations with social, diet-related, and neuropsychological factors. Nutrition. 2020 Mar;71:110640. doi: 10.1016/j.nut.2019.110640. Epub 2019 Nov 9. PMID 31812000
- [Background] Marcos-Delgado A, Yevenes-Briones H, Fernandez-Villa T, Martin-Sanchez V, Guallar-Castillon P, Rodriguez-Artalejo F, Lopez-Garcia E. Association between diet quality and malnutrition: pooled results from two population-based studies in older adults. BMC Geriatr. 2024 May 10;24(1):417. doi: 10.1186/s12877-024-04984-5. PMID 38730363
- [Background] Chen LK, Woo J, Assantachai P, Auyeung TW, Chou MY, Iijima K, Jang HC, Kang L, Kim M, Kim S, Kojima T, Kuzuya M, Lee JSW, Lee SY, Lee WJ, Lee Y, Liang CK, Lim JY, Lim WS, Peng LN, Sugimoto K, Tanaka T, Won CW, Yamada M, Zhang T, Akishita M, Arai H. Asian Working Group for Sarcopenia: 2019 Consensus Update on Sarcopenia Diagnosis and Treatment. J Am Med Dir Assoc. 2020 Mar;21(3):300-307.e2. doi: 10.1016/j.jamda.2019.12.012. Epub 2020 Feb 4. PMID 32033882
- [Background] Beckwee D, Delaere A, Aelbrecht S, Baert V, Beaudart C, Bruyere O, de Saint-Hubert M, Bautmans I. Exercise Interventions for the Prevention and Treatment of Sarcopenia. A Systematic Umbrella Review. J Nutr Health Aging. 2019;23(6):494-502. doi: 10.1007/s12603-019-1196-8. PMID 31233069
- [Background] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jan 1;48(1):16-31. doi: 10.1093/ageing/afy169. PMID 30312372
- [Background] Roubenoff R, Parise H, Payette HA, Abad LW, D'Agostino R, Jacques PF, Wilson PW, Dinarello CA, Harris TB. Cytokines, insulin-like growth factor 1, sarcopenia, and mortality in very old community-dwelling men and women: the Framingham Heart Study. Am J Med. 2003 Oct 15;115(6):429-35. doi: 10.1016/j.amjmed.2003.05.001. PMID 14563498
- [Background] Landi F, Cruz-Jentoft AJ, Liperoti R, Russo A, Giovannini S, Tosato M, Capoluongo E, Bernabei R, Onder G. Sarcopenia and mortality risk in frail older persons aged 80 years and older: results from ilSIRENTE study. Age Ageing. 2013 Mar;42(2):203-9. doi: 10.1093/ageing/afs194. Epub 2013 Jan 15. PMID 23321202